CLINICAL TRIAL: NCT04542304
Title: Efficacy of Diuretics in Kidney Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of resources
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Tammy Lisa Sirich, Assistant Professor of Medicine, Stanford University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 56566
Record Dates: First submitted 2020-08-27; First posted 2020-09-09 (Actual); Results first posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Chronic Kidney Disease; End Stage Renal Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic | interventions — Metolazone

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Metolazone then placebo (Active Comparator): Metolazone will be taken orally during the first week, followed by washout of 1-2 weeks, then placebo will be taken the following week.
  Interventions: Drug: Metolazone; Drug: Placebo
- Placebo then Metolazone (Placebo Comparator): Placebo will be taken orally during the first week, followed by washout of 1-2 weeks, then metolazone will be taken the following week.
  Interventions: Drug: Metolazone; Drug: Placebo

INTERVENTIONS:
Drug: Metolazone — Participants receive a single dose of metolazone.
Drug: Placebo — Participants receive a single dose of placebo to match metolazone.

SUMMARY:
This study will determine the efficacy of diuretics in patients with chronic kidney disease.

DETAILED DESCRIPTION:
Participants with chronic kidney disease will undergo two 1-week study periods (single-dose diuretic versus single-dose placebo) separated by 1-2 weeks of washout in a cross-over design. Blood and urine samples will be collected at the end of each study period to determine the effect on urine output and to assess the kidney clearance and levels of uremic solute. Participants will weigh themselves daily.

ELIGIBILITY:
Inclusion Criteria:

* stable chronic kidney disease patients able to provide consent
* stable dialysis patients who produce urine and able to provide consent

Exclusion Criteria:

* use of antibiotics for last two months or expected antibiotic use
* recent hospitalization or other event resulting in instability of food intake

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-06-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Stanford University, Palo Alto, California
  - VA Palo Alto Health Care System, Palo Alto, California

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 17 participants signed informed consent, and 6 were randomized to treatment.
Groups:
- Metolazone Then Placebo: Metolazone single dose taken orally during the first week, followed by washout of 1-2 weeks, then placebo single dose taken the following week.
- Placebo Then Metolazone: Placebo single dose taken orally during the first week, followed by washout of 1-2 weeks, then metolazone single dose taken the following week.
Period: Treatment Period 1 (1 Week)
Arm/Group | Metolazone Then Placebo | Placebo Then Metolazone
Started | 3 | 3
Completed | 3 | 3
Not Completed | 0 | 0
Period: Washout Period (2 Weeks)
Arm/Group | Metolazone Then Placebo | Placebo Then Metolazone
Started | 3 | 3
Completed | 3 | 3
Not Completed | 0 | 0
Period: Treatment Period 2 (1 Week)
Arm/Group | Metolazone Then Placebo | Placebo Then Metolazone
Started | 3 | 3
Completed | 3 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Metolazone Then Placebo | Placebo Then Metolazone | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (1.5) | 66 (13) | 66 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 2 | 3 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 2 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 0 | 0 | 0
  White | 2 | 1 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Change in Urine Output
Description: Average volume of urine produced in 24 hours.
Time Frame: Change from baseline urine output at 1 week for each study arm
Measure: Mean (Standard Deviation); unit: mL/day
Groups:
- Metolazone: Metolazone (single dose)
- Placebo: Placebo (single dose)
Arm/Group | Metolazone | Placebo
Number analyzed (Participants) | 6 | 6
mL/day | 809 (466) | 676 (487)

2. Secondary Outcome: Kidney Clearance of Uremic Solutes
Description: Kidney clearance of uremic solutes in ml/min.
Time Frame: Kidney clearance of uremic solutes at 1 week for each study arm
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Metolazone | Placebo
Number analyzed (Participants) | 6 | 6
mL/min
  P-Cresol sulfate | 15 (11) | 10 (8)
  Indoxyl sulfate | 34 (20) | 22 (15)
  Hippurate | 61 (48) | 42 (29)
  Phenylactyl glutamine | 14 (9) | 9 (7)

3. Secondary Outcome: Change in Quality of Life Questionnaire Score
Description: Kidney Disease Quality of Life 36 Questionnaire (KDQOL36)
Time Frame: Change from baseline quality of life score at 1 week for each study arm
Population: Because the plan was to administer the intervention as a single dose, the investigators determined that the KDQOL should be removed from the study design because it is an evaluation used to assess changes over time. This decision was made prior to enrollment of any participants and was not administered to any study participants; however, the measure was not removed from the registration at that time.
Arm/Group | Metolazone | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Plasma Urea
Time Frame: Week 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Metolazone | Placebo
Number analyzed (Participants) | 6 | 6
mg/dL | 54 (15) | 54 (13)

5. Secondary Outcome: Blood Pressure
Time Frame: Week 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Metolazone | Placebo
Number analyzed (Participants) | 6 | 6
mmHg
  Systolic | 140 (25) | 146 (18)
  Diastolic | 77 (13) | 76 (12)

6. Secondary Outcome: Weight Change
Time Frame: Baseline, Week 1
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Metolazone | Placebo
Number analyzed (Participants) | 6 | 6
kg
  Baseline | 74 (30) | 73 (31)
  Week 1 | 1.6 (1.7) | 1.9 (1.7)

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Metolazone | Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6

LIMITATIONS AND CAVEATS:
Early termination led to a small number of participants analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2023-03-15): https://cdn.clinicaltrials.gov/large-docs/04/NCT04542304/Prot_000.pdf
  • Statistical Analysis Plan (2025-04-14): https://cdn.clinicaltrials.gov/large-docs/04/NCT04542304/SAP_001.pdf